CLINICAL TRIAL: NCT05877807
Title: Effect of Baclofen to Prevent Post-Traumatic Stress Disorder: 5 Years Follow-up of the BACLOREA Randomized Trial
Brief Title: Effect of Baclofen to Prevent Post-Traumatic Stress Disorder
Acronym: BACLO-PTSD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0251
Record Dates: First submitted 2023-04-03; First posted 2023-05-26 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Alcoholism; Post Traumatic Stress Disorder
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Baclofen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental : BACLOFEN: Patient will receive baclofen caps
  Interventions: Drug: Baclofen
- Placebo Comparator : PLACEBO: Patient will receive placebo caps (lactose)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Baclofen — Daily doses will be adapted to daily MDRD creatinine clearance from 150 to 50mg. On the day of randomisation, the patient will receive the full daily dose in a one-shot administration. Then daily doses will be divided into 3 intakes on the following days. During the mechanical ventilation period, the treatment will be administered via the nasogastric feeding tube. After extubation, the treatment will be administered either via the nasogastric tube or the oral route.
  Groups: Experimental : BACLOFEN
Other: Placebo — Daily doses will be adapted to daily MDRD creatinine clearance from 150 to 50mg. On the day of randomisation, the patient will receive the full daily dose in a one-shot administration. Then daily doses will be divided into 3 intakes on the following days. During the mechanical ventilation period, the placebo will be administered via the nasogastric feeding tube. After extubation, the placebo will be administered either via the nasogastric tube or the oral route.
  Groups: Placebo Comparator : PLACEBO

SUMMARY:
Considering the results of the Baclorea study (10% reduction in episodes of agitation in intensive care in the Baclofen group), the investigators would like to know whether this reduction in agitation also results in a reduction in the incidence of the syndrome of long-term post-traumatic stress (5 years later).

The investigators wish to contact by telephone, blinded from the randomization group as defined in the framework of the Balorea project, by telephone contact, the patients who had been included in the Balorea study between June 2016 and February 2019.

DETAILED DESCRIPTION:
Background: Alcohol is the leading psychoactive substance consumed in France, with about 15 million regular consumers. The specific complication of alcoholism in the Intesive care is the alcohol withdrawal syndrome. Its incidence reaches up to 30% and its main complication is agitation. The Baclorea Randomized controlled Study showed that Baclofen significantly reduced the incidence of agitation in ICU but increased the length of stay in ICU. The BACLO-PTSD Study aims at assessing whether Baclofen administered during ICU stay to reduce the incidence of agitation could also reduce the incidence of Post-Traumatic Stress Disorder (PTSD) in mean term compared to placebo Methods/Design: This prospective, randomized, controlled study versus placebo will be conducted in eighteen French intensive care units (ICU). Patients included in the BACLO-REA Trial will have to respond to standardized questionnaires to detect Post-Traumatic Stress Disorder (Primary outcome) and to assess quality of life (Secondary outcome).

Discussion: Patients will be assessed blind to the randomization group. If patients in the Baclofen group present have a lower incidence of PTSD, the study will suggest that the increase in the length of ICU stay in the baclofen group could be beneficial to reduce the incidence of PTSD in patients with alcohol intake above de NIAAA recommendations.

ELIGIBILITY:
Inclusion Criteria :

All incident patients included in the BACLOREA trial. As a reminder, the criteria were :

* Patients under guardianship/guardianship at the time of initial inclusion or since the end of the Balorea study will not be contacted and therefore will not be analyzed in this research.Non-cerebrodamaged patients admitted to intensive care regardless of the causal pathology with:
* Consumption of alcohol qualified as "at risk" (For men aged 18 to 64: Consumption ≥ 14 drinks/week in the month preceding hospitalization; For men > 65 and women: Consumption > 7 drinks /week in the month preceding hospitalization).
* AND Intubated, ventilated with an expected duration of mechanical ventilation of at least 48 hours;
* AND Aged 18 to 80

Exclusion Criteria :

* Patients who died during the study or within 5 years of inclusion will not be included. Also, patients who withdrew their consent after inclusion in the Balorea study will not be included. Similarly, patients refusing to answer telephone questionnaires will not be included. Known deceased patients will not be contacted.
* Patients under guardianship/guardianship at the time of initial inclusion or since the end of the Balorea study will not be contacted and therefore will not be analyzed in this research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who took part in the Baclorea study between 2016 and 2019. This study assessed the benefit of treatment with baclofen for the prevention of agitation in intensive care during the period of mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Assessment of the incidence of post-traumatic stress syndrome using the Revised Event Impact Scale (IES-R) | 5 years post hospitalization
  It has 2 important dimensions for the diagnosis of post-traumatic stress disorder: repetitive memories and persistent avoidance. The questionnaire is composed of 22 items to which the patient must respond using a scale of 0 to 4 (0 = not at all / 1 = a little / 2 = moderately / 3 = good-fair / 4 = extremely).
  Incidence of Post traumatic stress disorder defined by a score greater or equal to 33.

SECONDARY OUTCOMES:
Evaluation of the quality of life using the questionnaire European Quality of Life-5 Dimensions (EQ-5D) | 5 years post hospitalization
  For each of the headings (Mobility, Autonomy, Daily Activities, Pain/Discomfort, Anxiety/Depression), the patient must indicate the statement that best describes his state of health today. 3 answers are proposed indicating the level of difficulty (1 = no difficulty / 2 = average difficulty / 3 = extreme difficulty).
  The maximum value is 3 (wich is the worst outcome) and the minimum is 1 (wich is the best outcome).
Health assessement with the Short Form (SF-36 Quiz) | 5 years post hospitalization
  This health-related quality of life scale is made up of 36 questions, divided into 8 dimensions: physical activity, life and relationships with others, physical pain, perceived general health, vitality, limitations due to mental/physical state and mental health. The patient must answer all the questions. A circling the number corresponding to the chosen answer. At the end, a score for each dimension of the SF-36 is calculated, varying from 0 to 100. A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health.
Screen for anxiety and depressive disorders with Hospital Anxiety and Depression scale (HAD Quiz) | 5 years post hospitalization
  It has 14 rated items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus allowing two scores to be obtained (maximum score for each score = 21 wich is the worst state).
Evaluation of the Posttraumatic stress disorder (PCL-S Quiz) | 5 years post hospitalization
  The scale is composed of 17 items corresponding to the 3 syndromes main causes of PTSD : Intrusion, overstimulation and avoidance.
  Each question is to be scored between 1 and 5 depending on the intensity and frequency of the symptoms. The higher the total score on this 85-point scale, the worse is severe the post-traumatic stress disorder.
Assessment of patient Habits | 5 years post hospitalization
  Interrogation about Tobacco, alcohol and drug consumption (yes/no; type of drug; amount)

CONTACTS AND LOCATIONS:
Overall Officials: Karim ASEHNOUNE, PU-PH, Principal Investigator — Nantes University Hospital
Locations (13):
- France (13):
  - Brest University Hospital, Brest, Finistère
  - Cornouaille Hospital, Quimper, Finistère
  - Montpellier University Hospital, Montpellier, Hérault
  - Rennes University Hospital, Rennes, Ile-et-Vilaine
  - Tours University Hospital, Tours, Indre-et-Loire
  - Nantes University Hospital, Nantes, Loire-Atlantique
  - Saint-Nazaire Hospital, Saint-Nazaire, Loire-Atlantique
  - Angers University Hospital, Angers, Maine-et-Loire
  - South Bretagne Hospital Center, Lorient, Morbihan
  - Le Mans University Hospital, Le Mans, Sarthe
  - Vendee Departmental Hospital, La Roche-sur-Yon, Vendee
  - Poitiers University Hospital, Poitiers, Vienne
  - Saint-Antoine Hospital (AP-HP), Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bouras M, Asehnoune K, Robert-Valli Y, Mahe PJ, Reignier J, Maamar A, Lacherade JC, Jonas M, Jung B, Ferrandiere M, Jaber S, Flet L, Moriconi M, Lasocki S, Smonig R, Guitton C, Ehrmann S, Rozec B, Volteau C, Vourc'h M; BACLOREA study group. Effect of high-dose baclofen on post-traumatic stress disorder symptoms five years after hospitalization among critically ill patients with unhealthy alcohol use. Sci Rep. 2026 Jan 8;16(1):1088. doi: 10.1038/s41598-025-27423-w. PMID 41507241